CLINICAL TRIAL: NCT03134963
Title: Cerebral Haemodynamic Changes During Cognitive Testing: a Functional Transcranial Doppler (fTCD) Study
Brief Title: Cerebral Haemodynamic Changes During Cognitive Testing: A fTCD Study
Status: Completed | Type: Observational
Sponsor: University of Leicester (Other)
Responsible Party: Sponsor
Other Study IDs: 0613
Record Dates: First submitted 2017-03-09; First posted 2017-05-01 (Actual); Results first posted 2020-11-25 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2017-03

CONDITIONS: Mild Cognitive Impairment; Alzheimer Disease; Vascular Dementia; Healthy Controls
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Dementia, Vascular | interventions — Ultrasonography, Doppler, Transcranial; Blood Pressure Monitors

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Mild cognitive impairment: MCI Patient-specific Inclusion Criteria
  Clinical diagnosis of MCI made by a specialist* in a patient who fulfils the established clinical consensus criteria for MCI [NIA/AA 2011] specifically:
  * Concern regarding a change in cognition compared to the person's previous level, by the patient and/or informant
  * Objective evidence of impairment of one or more cognitive domains, greater than expected for age, and educational background, over time if repeated measures are available.
  * Preserved independence of functional abilities and minimal to no impairment on complex instrumental functions
  * Not demented
  Interventions: Other: Transcranial doppler ultrasonography; Other: Blood pressure monitoring; Other: Heart rate monitoring; Other: End tidal CO2 monitoring; Other: Addenbrooke's cognitive examination
- Alzheimer disease: NIA/AA criteria
  * Meets the criteria for dementia
    o The memory impairment and cognitive deficits cause significant impairment functioning, a significant decline from a previous level of functioning, Impairment of at least two cognitive domains
  * Insidious or gradual onset
  * Clear history of worsening cognition by report or observation
  * The initial and most prominent cognitive deficits are evident on history and examination in one of the following domains:
    * Amnestic: impaired learning and recall of recently learned information
    * Non amnestic: language/visuospatial/executive dysfunction
  Interventions: Other: Transcranial doppler ultrasonography; Other: Blood pressure monitoring; Other: Heart rate monitoring; Other: End tidal CO2 monitoring; Other: Addenbrooke's cognitive examination
- Vascular dementia: NINDS-AIREN criteria for VascD, specifically:
  * Cerebrovascular disease defined by the presence of focal signs on neurological examination consistent with stroke and evidence of cerebrovascular disease on brain imaging.
  * One or more of:
    * Onset of dementia within 3 months of a diagnosed stroke
    * Abrupt deterioration in cognitive function
    * Fluctuating, stepwise progression of cognitive deficits
  Interventions: Other: Transcranial doppler ultrasonography; Other: Blood pressure monitoring; Other: Heart rate monitoring; Other: End tidal CO2 monitoring; Other: Addenbrooke's cognitive examination
- Healthy controls: Healthy Controls-specific Inclusion Criteria
  1. No evidence of subjective or objective memory impairment on cognitive testing
  2. No major medical co-morbidity (outlined in detail in the exclusion criteria) or medication use that could adversely affect cognition
  Interventions: Other: Transcranial doppler ultrasonography; Other: Blood pressure monitoring; Other: Heart rate monitoring; Other: End tidal CO2 monitoring; Other: Addenbrooke's cognitive examination

INTERVENTIONS:
Other: Transcranial doppler ultrasonography — Measurement of cerebral blood flow whilst undertaking cognitive tasks with TCD monitoring.
  Other Names: TCD
Other: Blood pressure monitoring — Continuous blood pressure recording
  Other Names: Finometer
Other: Heart rate monitoring — Continuous heart rate monitoring
  Other Names: Electrocardiogram
Other: End tidal CO2 monitoring — Continuous ETCO2 monitoring
  Other Names: Capnography
Other: Addenbrooke's cognitive examination — Performance of a memory test
  Other Names: ACE III

SUMMARY:
850,000 people live with dementia in the UK, with that number expected to rise to more than 1 million within the next 5 years. The most common type of dementia (55%) is Alzheimer's dementia, and vascular dementia is the second commonest type (15%). Mild cognitive impairment (MCI) affects up to 20% of older adults and describes a set of symptoms rather than a specific medical condition or disease. A person with MCI has subtle problems with one or more of the following: day-to-day memory, concentrating, planning or organising, language (eg struggling to find the right word), and judging distances and seeing objects properly. Although MCI significantly increases the risk of developing dementia (by up to 5 times), at present it is not possible to accurately predict which patients with MCI will progress to dementia. In recent times there has been an increasing awareness that problems with brain blood flow may contribute to the development, or progression, of dementia. Tests of mental abilities, with standardised questions and pen-and-paper tests are a key component of the formal diagnosis of dementia, yet little is known of the effects of these tests on brain blood flow. Brain blood flow can be can be assessed non-invasively by the use of Trans Cranial Doppler (TCD). This means using ultrasound probes over both sides of the head to measure changes in blood flow in one of the main brain arteries (the middle cerebral artery). This proposed study will therefore use TCD to evaluate changes in brain blood flow during performance of the Addenbrooke's-III (ACE-III) cognitive assessment in four key groups of patients, specifically:

1. Healthy older adults
2. Patients with mild cognitive impairment (MCI)
3. Patients with vascular dementia
4. Patients with Alzheimer's dementia

DETAILED DESCRIPTION:
Dementia is the most common neurodegenerative disorder in the United Kingdom (UK); 850,000 people currently live with dementia in the UK, and that number is expected to rise to more than 1 million within the next 5 years. The annual cost to the UK of dementia is £23.6 billion. The most common type of dementia in the population (55%) is Alzheimer's dementia (AlzD). AlzD typically has a gradual onset and a slow progression. Vascular dementia (VascD) is the second commonest form of dementia (15%), and is suggested by the presence of vascular risk factors such as high blood pressure, high cholesterol, smoking and heart disease. The onset of vascular dementia is often abrupt, and the progression stepwise and irregular; cognitive deficits are often less uniform than those of Alzheimer's dementia. Mild cognitive impairment (MCI) affects up to 20% of older adults and describes a set of symptoms rather than a specific medical condition or disease. A person with MCI has subtle problems with one or more of the following: day-to-day memory, planning, language, attention and visuospatial skills. Although MCI significantly increases the risk of developing dementia at present it is not possible to accurately predict which patients with MCI will progress to dementia.

In recent times, our knowledge regarding the mechanisms of dementia development has changed considerably. In contrast to previous thoughts, there is now a growing understanding that problems with blood vessels (vascular dysfunction) and brain blood flow (cerebral haemodynamics) are present in AlzD as well as in VascD. Research studies investigating the vascular contributions to dementia generally report low blood flow (cerebral hypoperfusion). It is thought that this hypoperfusion affects cellular health which in turn triggers neurodegenerative pathways.

Brain blood flow is directly linked to brain activity, a concept known as 'neurovascular coupling'. Brain activation can be achieved through various cognitive and visual tasks (e.g reading and writing), and also by sensorimotor tasks (e.g. movement or touch). Cognitive assessments are routinely used in the diagnosis of dementia. Brain blood flow can be studied using techniques such as functional magnetic resonance imaging (fMRI), positron emission tomography (PET) or single-photon emission computed tomography (SPECT). However, these techniques are expensive, in the case of SPECT involve radiation, and there are feasibility issues which are particularly problematic for older populations, including the need to lie still for prolonged periods and have no metal implants. Transcranial Doppler (TCD) ultrasound is a simple, non-invasive imaging technique which allows for the continuous and bilateral recording of brain blood flow velocity through the major arteries in the brain.

Cognitive testing with standardised assessment tools such as the Mini Mental State Examination, Montreal Cognitive Assessment and Addenbrooke's-III Cognitive Examination (ACE-III) is a key component of the formal diagnosis of dementia, yet the effects of these tests on brain blood flow and haemodynamics is unknown. The ACE-III is a widely used, validated, cognitive screening tool recommended for use by health practitioners and researchers in patients over 50 years old with suspected dementia. The ACE-III is available for free. The copyright is held by Professor John Hodges, ARC Federation Fellow and Professor of Cognitive Neurology at Neuroscience Research Australia, who is happy for the test to be used in clinical practice and research projects.

This protocol has been used successfully by this group to examine changes in CBFv in 40 healthy volunteers from the University of Leicester. The data from this analysis has been presented at an international conference and is currently undergoing peer review for publication. Therefore, this protocol has demonstrated feasibility in a healthy population and warrants further investigation for the utility in a patient population.

This research will therefore use transcranial Doppler ultrasound to study the brain blood flow responses of healthy controls, patients with AlzD, patients with VascD, and patients with MCI, in response to performance of the ACE-III cognitive examination.

ELIGIBILITY:
Inclusion Criteria:

* Informed volunteer consent, patient consent
* Male or female, aged between 18 and 100 years of age
* Able (in the Investigator's opinion) and willing to comply with all study requirements
* Willing to allow his or her General Practitioner (GP) to be notified of participation in the study
* Good understanding of written and verbal English

Healthy Controls-specific Inclusion Criteria

* No evidence of subjective or objective memory impairment on cognitive testing
* No major medical co-morbidity (outlined in detail in the exclusion criteria) or medication use that could adversely affect cognition

MCI Patient-specific Inclusion Criteria

Clinical diagnosis of MCI made by a specialist* in a patient who fulfils the established clinical consensus criteria for MCI [NIA/AA 2011] specifically:

* Concern regarding a change in cognition compared to the person's previous level, by the patient and/or informant
* Objective evidence of impairment of one or more cognitive domains, greater than expected for age, and educational background, over time if repeated measures are available.
* Preserved independence of functional abilities and minimal to no impairment on complex instrumental functions
* Not demented

Vascular Dementia Specific Inclusion Criteria

Clinical diagnosis of VascD made by a specialist* in a patient who fulfils the NINDS-AIREN criteria for VascD, specifically:

* Cerebrovascular disease defined by the presence of focal signs on neurological examination consistent with stroke and evidence of cerebrovascular disease on brain imaging.
* One or more of:

  * Onset of dementia within 3 months of a diagnosed stroke
  * Abrupt deterioration in cognitive function
  * Fluctuating, stepwise progression of cognitive deficits

Alzheimer's Dementia Specific Inclusion Criteria

Clinical Diagnosis of AlzD made by a specialist* in a patient who fulfils the NIA/AA criteria for Probable AlzD, specifically:

* Meets the criteria for dementia

  * The memory impairment and cognitive deficits cause significant impairment in social or occupational functioning, and represent a significant decline from a previous level of functioning, not explained by a delirium or a major psychiatric disorder
  * Impairment of at least two cognitive domains
* Insidious or gradual onset
* Clear history of worsening cognition by report or observation
* The initial and most prominent cognitive deficits are evident on history and examination in one of the following domains:

  * Amnestic: impaired learning and recall of recently learned information
  * Non amnestic: language/visuospatial/executive dysfunction
* No evidence of substantial cerebrovascular disease, core features of dementia with lewy bodies, features of frontotemporal dementia, prominent features of semantic variant primary progressive aphasia, evidence of active neurological disease, a non-neurological co-morbidity or medication that could affect cognition

  * A specialist being defined as a psychiatrist or a geriatrician, or a specialist mental health nurse with a specific interest or expertise in cognitive disorders.

Exclusion Criteria:

Exclusion Criteria

* Male or Female, aged under 18 years
* Unable (in the Investigator's opinion) or unwilling to comply with any study requirements
* Female participants who are pregnant, lactating or planning pregnancy during the course of the study
* Major co-morbidity likely to affect cerebral autoregulation; severe respiratory disease, carotid artery stenosis, atrial fibrillation, severe cardiac failure (left ventricular ejection fraction <20%), extreme frailty or multi-morbidity.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy controls - age, sex and co-morbidity matched. Patients with Alzheimer's dementia, vascular dementia, and mild cognitive impairment
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2017-05-05 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thompson G Robinson, MD, Principal Investigator — University of Leicester
Locations (2):
- United Kingdom (2):
  - University Hospitals of Leicester NHS Trust, Leicester, Leicestershire
  - Leicestershire Partnership Trust, Leicester, Leicestershire

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Mild Cognitive Impairment: MCI Patient-specific Inclusion Criteria
  Clinical diagnosis of MCI made by a specialist* in a patient who fulfils the established clinical consensus criteria for MCI [NIA/AA 2011] specifically:
  * Concern regarding a change in cognition compared to the person's previous level, by the patient and/or informant
  * Objective evidence of impairment of one or more cognitive domains, greater than expected for age, and educational background, over time if repeated measures are available.
  * Preserved independence of functional abilities and minimal to no impairment on complex instrumental functions
  * Not demented
  Transcranial doppler ultrasonography: Measurement of cerebral blood flow whilst undertaking cognitive tasks with TCD monitoring.
  Blood pressure monitoring: Continuous blood pressure recording
  Heart rate monitoring: Continuous heart rate monitoring
  End tidal CO2 monitoring: Continuous ETCO2 monitoring
  Addenbrooke's cognitive examination: Performance of a memory test
- Alzheimer Disease: NIA/AA criteria
  * Meets the criteria for dementia
    o The memory impairment and cognitive deficits cause significant impairment functioning, a significant decline from a previous level of functioning, Impairment of at least two cognitive domains
  * Insidious or gradual onset
  * Clear history of worsening cognition by report or observation
  * The initial and most prominent cognitive deficits are evident on history and examination in one of the following domains:
    * Amnestic: impaired learning and recall of recently learned information
    * Non amnestic: language/visuospatial/executive dysfunction
  Transcranial doppler ultrasonography: Measurement of cerebral blood flow whilst undertaking cognitive tasks with TCD monitoring.
  Blood pressure monitoring: Continuous blood pressure recording
  Heart rate monitoring: Continuous heart rate monitoring
  End tidal CO2 monitoring: Continuous ETCO2 monitoring
  Addenbrooke's cognitive examination: Performance of a memory test
- Vascular Dementia: NINDS-AIREN criteria for VascD, specifically:
  * Cerebrovascular disease defined by the presence of focal signs on neurological examination consistent with stroke and evidence of cerebrovascular disease on brain imaging.
  * One or more of:
    * Onset of dementia within 3 months of a diagnosed stroke
    * Abrupt deterioration in cognitive function
    * Fluctuating, stepwise progression of cognitive deficits
  Transcranial doppler ultrasonography: Measurement of cerebral blood flow whilst undertaking cognitive tasks with TCD monitoring.
  Blood pressure monitoring: Continuous blood pressure recording
  Heart rate monitoring: Continuous heart rate monitoring
  End tidal CO2 monitoring: Continuous ETCO2 monitoring
  Addenbrooke's cognitive examination: Performance of a memory test
- Healthy Controls: Healthy Controls-specific Inclusion Criteria
  1. No evidence of subjective or objective memory impairment on cognitive testing
  2. No major medical co-morbidity (outlined in detail in the exclusion criteria) or medication use that could adversely affect cognition
  Transcranial doppler ultrasonography: Measurement of cerebral blood flow whilst undertaking cognitive tasks with TCD monitoring.
  Blood pressure monitoring: Continuous blood pressure recording
  Heart rate monitoring: Continuous heart rate monitoring
  End tidal CO2 monitoring: Continuous ETCO2 monitoring
  Addenbrooke's cognitive examination: Performance of a memory test
Period: Overall Study
Arm/Group | Mild Cognitive Impairment | Alzheimer Disease | Vascular Dementia | Healthy Controls
Started | 12 | 13 | 3 | 14
Completed | 12 | 13 | 3 | 14
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mild Cognitive Impairment | Alzheimer Disease | Vascular Dementia | Healthy Controls | Total
Number analyzed (Participants) | 12 | 13 | 3 | 14 | 42
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 72 [70 to 79.5] | 76 [72 to 82] | 83 [83 to 83] | 71 [64.5 to 74] | 73.5 [70.25 to 78.25]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 0 | 4 | 10
  Male | 9 | 10 | 3 | 10 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 13 | 3 | 14 | 42
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Recruited Subjects Able to Comply With the Protocol
Description: The percentage of recruited subjects (HC, MCI patients, VascD patients and AlzD patients) able to comply with the full measurement protocol.
Time Frame: 8 months
Measure: Count of Participants; unit: Participants
Arm/Group | Mild Cognitive Impairment | Alzheimer Disease | Vascular Dementia | Healthy Controls
Number analyzed (Participants) | 12 | 13 | 3 | 14
Participants | 12 | 13 | 3 | 14

2. Secondary Outcome: Number of Participants With Rejected Measurements
Description: The percentage of measurements rejected because of aspects related to data quality during the analysis protocol, with recorded reasons
Time Frame: 8 months
Measure: Count of Participants; unit: Participants
Arm/Group | Mild Cognitive Impairment | Alzheimer Disease | Vascular Dementia | Healthy Controls
Number analyzed (Participants) | 12 | 13 | 3 | 14
Participants | 2 | 3 | 0 | 4

3. Secondary Outcome: Number of Participants in Which Percentage Change in CBFv Can be Derived
Description: Overall, the percentage of recruited subjects (healthy controls, MCI patients, VascD patients and AlzD patients) in whom values for the following parameters can be derived:
  • % change of CBFv at baseline in response to performance of the ACE-III Cognitive Examination
Time Frame: 8 months
Measure: Count of Participants; unit: Participants
Arm/Group | Mild Cognitive Impairment | Alzheimer Disease | Vascular Dementia | Healthy Controls
Number analyzed (Participants) | 12 | 13 | 3 | 14
Participants | 10 | 10 | 3 | 10

4. Secondary Outcome: Number of Participants in Which the Change in the Autoregulation Index (ARI) Can be Derived
Description: Overall, the percentage of recruited subjects (healthy controls, MCI patients, VascD patients and AlzD patients) in whom values for the following parameters can be derived:
  • Autoregulation index (using the Tiecks model and from the phase, gain and coherence).
Time Frame: 8 months
Measure: Count of Participants; unit: Participants
Arm/Group | Mild Cognitive Impairment | Alzheimer Disease | Vascular Dementia | Healthy Controls
Number analyzed (Participants) | 12 | 13 | 3 | 14
Participants | 10 | 10 | 3 | 10

ADVERSE EVENTS:
Time Frame: 3 months
Description: Definition: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Arm/Group | Mild Cognitive Impairment | Alzheimer Disease | Vascular Dementia | Healthy Controls
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/13 | 0/3 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/13 | 0/3 | 0/14
Other Adverse Events (participants affected / at risk) | 0/12 | 0/13 | 0/3 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-01): https://cdn.clinicaltrials.gov/large-docs/63/NCT03134963/Prot_SAP_000.pdf